CLINICAL TRIAL: NCT03764826
Title: Study on the Effect of Sound Therapy on Chronic Primary Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Shu-sheng Gong, director of Department of Otorhinolaryngology Head and Neck Surgery, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-P2-182-01
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAABT (Experimental): CAABT(Cochleural Alternating Acoustic Beam Therapy) is an innovative tinnitus intervention which based on neural science and cochlear plastic research and aimed to reprogram the central auditory system to neutralize the discordant responses of the dysfunctioning cochlea via acoustic beaming stimuli.
  Interventions: Device: CAABT
- TMT (Active Comparator): TMT(tinnitus masking therapy) is a traditional tinnitus intervention. The masking sound is mainly white noise, and the intensity just covers tinnitus.
  Interventions: Device: TMT

INTERVENTIONS:
Device: CAABT — The sound generators with CAABT will be used 15 min each session, three times a day
  Arms: CAABT
Device: TMT — The sound generators with TMT will be used 15 min each session, three times a day
  Arms: TMT

SUMMARY:
This study is to compare the effect of Cochleural Alternating Acoustic Beam Therapy(CAABT) and tinnitus masking therapy(TMT) on chronic primary tinnitus.Half of participants will receive CAABT, while the other half will receive TMT.

DETAILED DESCRIPTION:
The patients with tinnitus will be collected with medical history, ear examination ,auditory function test and questionnaire survey.100 cases of chronic primary tinnitus will be selected as the research object.This study will be developed in the form of a blind randomized clinical trial.The study subjects will be divided into 2 groups by randomized method, with 50 cases in each group. Psychological acoustic test, Resting-state function magnetic resonance imaging（RS-fMRI) will be conducted.For 6 months, the patients will be treated with Cochleural Alternating Acoustic Beam Therapy（CAABT）and tinnitus masking therapy（TMT） respectively, followed by questionnaire survey, psychological acoustics test and RS-fMRI. The THI,VAS score, RS-fMRI ReHo value and low-frequency wave amplitude (ALFF) before and after the treatment will be compared. For those cases with poor results, the exchanged treatment will be performed for 6 months, followed by questionnaire survey, psychoacoustic test, RS-fMRI, and comparison of THI, VAS score, ReHo value and ALFF before and after treatment.All cases will be followed up for 1 year, and questionnaire survey will be conducted again.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-75 years
* Tinnitus undergone for more than 6 months
* Continuous attack, single tone dominated, annoying tinnitus
* Able to cooperate with auditory function test and psychoacoustic test
* The main tinnitus frequency is from 125Hz to 8000Hz
* Willing to use the equipment daily during the test
* Willing and able to follow up regularly
* Ability to read and write Chinese, able to understand and complete questionnaires

Exclusion Criteria:

* Secondary tinnitus
* Pure tone audiometry shows conduction deafness or mixed deafness
* Tinnitus main frequency threshold >60dB
* Receiving treatment for other tinnitus
* MRI contraindications
* Feeling uncomfortable with the treatment equipment or not being accepted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-08 (Estimated); Study Completion 2019-12-08 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory ( THI) | baseline, 2 months, 4 months, 6 months
  Change from Baseline in Tinnitus Subjective Measures at 2 months, 4 months, 6 months: Tinnitus Handicap Inventory scale.
  Efficacy evaluation criteria: (1) cure: THI score was reduced to less than 16 points;(2) significant effect: THI score decreased by more than 17 points;(3) invalid: THI score value decreased < 17 points or even increased.Efficiency is the sum of cure and effect.
Resting-state function magnetic resonance imaging(RS-fMRI) Regional homogeneity(ReHo) value | baseline, 6 months
  Change from Baseline in Tinnitus Subjective Measures at 6 months: RS-fMRI ReHo value
Resting-state function magnetic resonance imaging(RS-fMRI) low-frequency wave amplitude (ALFF) | baseline, 6 months
  Change from Baseline in Tinnitus Subjective Measures at 6 months: RS-fMRI ALFF
Visual Analogue Scale(VAS) | baseline, 2 months, 4 months, 6 months
  Change from Baseline in Tinnitus Subjective Measures at 2 months, 4 months, 6 months: Visual Analogue Scale(VAS).
  The number 0 to 10 indicates the severity of symptoms, "0" means no symptoms, and "10" means the most severe

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Sheng Gong, MD, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available within 6 months of study completion
Supporting Information: Study Protocol
Time Frame: Data access requests will be reviewed by an external Independent Review Panel.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel

REFERENCES:
- [Result] Tunkel DE, Bauer CA, Sun GH, Rosenfeld RM, Chandrasekhar SS, Cunningham ER Jr, Archer SM, Blakley BW, Carter JM, Granieri EC, Henry JA, Hollingsworth D, Khan FA, Mitchell S, Monfared A, Newman CW, Omole FS, Phillips CD, Robinson SK, Taw MB, Tyler RS, Waguespack R, Whamond EJ. Clinical practice guideline: tinnitus executive summary. Otolaryngol Head Neck Surg. 2014 Oct;151(4):533-41. doi: 10.1177/0194599814547475. PMID 25274374
- [Result] Liu C, Lv H, Jiang T, Xie J, He L, Wang G, Liu J, Wang Z, Gong S. The Cochleural Alternating Acoustic Beam Therapy (CAABT): A pre-clinical trial. Am J Otolaryngol. 2018 Jul-Aug;39(4):401-409. doi: 10.1016/j.amjoto.2018.04.002. Epub 2018 Apr 3. PMID 29655489